CLINICAL TRIAL: NCT00034749
Title: The Efficacy and Safety of Risperidone in Adolescents With Schizophrenia: a Comparison of Two Dose Ranges of Risperidone
Brief Title: The Efficacy and Safety of Risperidone in the Treatment of Adolescents With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003361
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Adolescents; Schizophrenia; risperidone
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
A clinical study to compare the safety and effectiveness of two different dose ranges of risperidone solution in the treatment of adolescents with a diagnosis of schizophrenia.

DETAILED DESCRIPTION:
This is a clinical study of an investigational drug called risperidone in the treatment of schizophrenia in adolescents. Initially children (age 2 to 12 yrs) and schizophreniform subjects were also allowed but excluded following protocol amendment.

The study will include approximately 260 patients aged 13 to 17 years with a diagnosis of schizophrenia. Subjects will be randomly assigned to one of two groups on enrollment and will be given risperidone as an oral solution each day for 8 weeks at doses within one of two dose different ranges, according to the assigned study group.

Initially the two dose range were 0.15-0.4 mg/day and 1.5-4mg/day but were changed in protocol amendment to evaluate the maximum tolerated dose with a minimum of 3.5mg/day and maximum of 6mg/day (resp. 0.35 and 0.6mg/day in low dose treatment arm) Risperidone lower dose (0.35-0.6 mg/day [subjects >=50kg] or 0.007-0.012 mg/kg/day [subjects <50 kg]) as 0.1 mg/mL oral solution or risperidone higher dose (3.5-6 mg/day [subjects >=50 kg] or 0.07-0.12 mg/kg/day [subjects <50 kg]) as 1 mg/mL oral solution for 8 weeks. Daily dose can be given all at once or through 2 administrations (in morning and evening); the dose is increased based on efficacy and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible for study enrollment if they: are adolescents between the ages of 13 and 17 years
* have a confirmed diagnosis of schizophrenia and are suffering from an acute episode
* provide their assent and parental informed consent to participate
* are otherwise relatively healthy on the basis of a medical and physical examination
* and are able to be in-patients for approximately 2 weeks.

Exclusion Criteria:

* Subjects will be excluded from the study if they: meet the criteria for psychiatric disorders other than schizophrenia
* have moderate or severe mental retardation
* fail to respond to treatment with at least two typical or atypical antipsychotics
* have a history of substance dependence within the 3 months before screening
* are considered at risk for suicidal or violent behavior
* have a seizure disorder
* have a history of neuroleptic malignant syndrome, similar encephalopathic syndrome, or tardive dyskinesia
* or receive prohibited medication within a specified period before screening.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 279 (Actual)
Dates: Start 2001-04; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Change in total PANSS (Positive and Negative Syndrome Scale for Schizophrenia) from baseline to the 8-week endpoint

SECONDARY OUTCOMES:
Change from baseline in PANSS subscale scores and Clinical Global Impression (CGI-S and CGI-I) scores, number of subjects achieving a clinical response (at least 20% improvement in total PANSS), safety, tolerability and pharmacokinetics.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Haas M, Eerdekens M, Kushner S, Singer J, Augustyns I, Quiroz J, Pandina G, Kusumakar V. Efficacy, safety and tolerability of two dosing regimens in adolescent schizophrenia: double-blind study. Br J Psychiatry. 2009 Feb;194(2):158-64. doi: 10.1192/bjp.bp.107.046177. PMID 19182179
- See also: The Efficacy and Safety of Risperidone in the Treatment of Adolescents With Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=521&filename=CR003361_CSR.pdf